CLINICAL TRIAL: NCT07267377
Title: Effects of Sedation Techniques on Early Cognitive Recovery in Ambulatory Gynecologic Surgery: A Prospective Randomized Study
Brief Title: Effects of Different Sedation Techniques on Early Cognitive Recovery After Ambulatory Gynecologic Surgery
Acronym: SEDCOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sait Fatih Öner (Other)
Responsible Party: Sponsor-Investigator, Sait Fatih Öner, Principal Investigator, Elazıg Fethi Sekin Sehir Hastanesi
Organization: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: no.258551508; November 5, 2024; no.258551508; November 5, 2024 (Other: Elazig Fethi Sekin City Hospital Ethics Committee)
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Recovery; Sedation; Ambulatory Gynecologic Surgery; Postoperative Recovery
Keywords: Propofol; Ketamine; Ketofol; Sedoanalgesia; Cognitive Recovery; Ambulatory Surgery; Gynecologic Surgery; Postoperative Recovery; Mini-Mental State Examination
MeSH Terms: interventions — Propofol; Fentanyl; Ketamine

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model with three groups of participants. Each group receives a different sedoanalgesic regimen: propofol-fentanyl, ketamine-fentanyl, or propofol + ketamine + fentanyl (ketofol).
  Outcomes related to early cognitive recovery and hemodynamic stability are compared among the groups.
Who Masked: Participant, Investigator
Masking Description: Both the participants and the investigators administering sedation were blinded to the group assignments.
  Sedative solutions were prepared in identical syringes by an independent anesthesiologist not involved in data collection or analysis.
  The assessing investigator was unaware of the sedative regimen used for each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol-Fentanyl Group (Active Comparator): Induction propofol 0.5 mg/kg + fentanyl 1 µg/kg; maintenance propofol 0.25 mg/kg as intermittent boluses to maintain RSS=3
  Interventions: Drug: Propofol-Fentanyl
- Ketamine-Fentanyl Group (Active Comparator): Induction ketamine 0.5 mg/kg + fentanyl 1 µg/kg; maintenance ketamine 0.25 mg/kg as intermittent boluses
  Interventions: Drug: Ketamine-Fentanyl
- Propofol + Ketamine + Fentanyl Group (Ketofol) (Active Comparator): Induction ketofol 0.75 mg/kg (1:1 mixture of propofol 10 mg/mL and ketamine 50 mg/mL, freshly prepared in a single syringe) + fentanyl 1 µg/kg; maintenance ketofol 0.25 mg/kg as intermittent boluses
  Interventions: Drug: Propofol + Ketamine + Fentanyl (Ketofol)

INTERVENTIONS:
Drug: Propofol-Fentanyl — Intravenous administration of propofol 0.5 mg/kg + fentanyl 1 µg/kg for sedation during ambulatory dilation and curettage (D&C).
  This regimen represents the standard sedoanalgesia practice for gynecologic day-case procedures and serves as one of the comparison arms in the study.
  Other Names: Propofol (Diprivan); Fentanyl (Fentanyl Citrate)
  Arms: Propofol-Fentanyl Group
Drug: Ketamine-Fentanyl — Intravenous administration of ketamine 0.5 mg/kg + fentanyl 1 µg/kg for sedation during ambulatory dilation and curettage (D&C).
  This arm evaluates the effects of ketamine-based sedoanalgesia on cognitive and hemodynamic recovery compared with other regimens.
  Other Names: Ketamine (Ketalar) Fentanyl (Fentanyl Citrate)
  Arms: Ketamine-Fentanyl Group
Drug: Propofol + Ketamine + Fentanyl (Ketofol) — Intravenous co-administration of propofol 0.5 mg/kg, ketamine (0.5 mg/kg), and fentanyl (1 µg/kg) for sedation during ambulatory dilation and curettage (D&C).
  This combination (known as "Ketofol") aims to balance the sedative and hemodynamic effects of propofol and ketamine, and is compared with single-agent sedoanalgesia regimens.
  Other Names: Propofol (Diprivan) Ketamine (Ketalar) Fentanyl (Fentanyl Citrate)
  Arms: Propofol + Ketamine + Fentanyl Group (Ketofol)

SUMMARY:
This prospective, randomized, double-blind clinical trial aims to compare the effects of three commonly used sedoanalgesia regimens on early cognitive recovery in patients undergoing ambulatory gynecologic surgery (dilatation and curettage).

The main objective of the study is to determine whether the use of propofol-fentanyl, ketamine-fentanyl, or their combination (ketofol-fentanyl) influences the recovery of cognitive functions during the early postoperative period.

The primary outcome is the change in the Mini-Mental State Examination (MMSE) score between baseline and recovery.

Secondary outcomes include awakening time, Aldrete recovery score (ARS), pain intensity using the visual analog scale (VAS) at 10 and 30 minutes, hemodynamic parameters, and adverse events.

Participants will be randomly assigned to one of three groups:

Group P: Propofol-fentanyl

Group K: Ketamine-fentanyl

Group KP: Propofol + ketamine + fentanyl

All patients will receive sedation to achieve a Ramsay Sedation Scale score of 3-4. Cognitive function will be assessed preoperatively and after recovery in the post-anesthesia care unit.

The study seeks to determine whether the combined use of ketamine and propofol provides any advantage in cognitive recovery or hemodynamic stability compared to single-agent sedation.

DETAILED DESCRIPTION:
Early postoperative cognitive recovery is an important indicator of patient safety and discharge readiness in ambulatory anesthesia. Various sedative-analgesic combinations are used for gynecologic day-case procedures; however, their effects on early cognitive recovery remain unclear.

This prospective, randomized, double-blind clinical trial was conducted to compare the effects of three commonly used sedoanalgesia regimens - propofol-fentanyl, ketamine-fentanyl, and their combination (ketofol-fentanyl) - on postoperative cognitive function recovery after dilation and curettage (D&C).

A total of 108 ASA physical status I-III patients aged 18-60 years were included and randomly allocated into three groups (n=36 each). Sedation was titrated to maintain a Ramsay Sedation Scale (RSS) score of 3-4. Cognitive function was assessed preoperatively and postoperatively using the Mini-Mental State Examination (MMSE).

The primary outcome was the change in MMSE score between baseline and recovery. Secondary outcomes included awakening time, Aldrete recovery score (ADS), visual analog scale (VAS) pain score at 10 and 30 minutes, hemodynamic stability, and adverse events.

The study aimed to identify the sedative regimen that optimizes cognitive recovery and minimizes side effects in ambulatory gynecologic anesthesia, contributing to safer and faster discharge decisions.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-60 years
* ASA physical status I-III
* Scheduled for ambulatory dilation and curettage (D&C) under sedoanalgesia
* No neurological or psychiatric disorders

Exclusion Criteria:

* History of neurological, psychiatric, or cognitive disorders
* Inability to complete or comprehend cognitive assessment tests (MMSE)
* Known drug or alcohol abuse
* Pregnancy
* Severe hepatic or renal dysfunction

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Mini-Mental State Examination (MMSE) Score | Baseline and recovery (within approximately 60 minutes post-sedation)
  Difference between baseline and postoperative MMSE scores measured before sedation and at recovery in the post-anesthesia care unit (PACU). The MMSE assesses early cognitive recovery after ambulatory gynecologic surgery under sedation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fethi Sekin City Hospital, Elâzığ, Elaziğ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study was conducted as a prospective, randomized, double-blind clinical trial at a single center.
  Individual participant data (IPD) will not be shared because no consent for data sharing beyond the study team was obtained, and there is no approved external repository for data storage